CLINICAL TRIAL: NCT04368351
Title: Evaluation of the Impact of Bacteriotherapy in the Treatment of COVID-19
Brief Title: Bacteriotherapy in the Treatment of COVID-19
Acronym: BACT-ovid
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giancarlo Ceccarelli, MD, PhD, MSc, University of Roma La Sapienza
Other Study IDs: DPHID-UniRoma05
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: COVID; Pneumonia; Diarrhea
Keywords: COVID-19 pneumonia; gut-lung axis; microbiome
MeSH Terms: conditions — Pneumonia; Diarrhea | interventions — Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of care: Azithromycin 500mg 1 cp / day (alternatively lopinavir/ritonavir cps 200/50 mg, 2 cps x 2 / day or darunavir 800 mg 1 cp / day + ritonavir 100 mg 1 cp / day or darunavir/cobicistat 800/150 mg 1 cp / day), plus hydroxychloroquine cp 200 mg, 1 cp x 2 / day.
  Interventions: Drug: Azithromycin; Drug: hydroxychloroquine
- bacteriotherapy: Dietary Supplement: SivoMixx (200 billion) plus Azithromycin 500mg 1 cp / day (alternatively lopinavir/ritonavir cps 200/50 mg, 2 cps x 2 / day or darunavir 800 mg 1 cp / day + ritonavir 100 mg 1 cp / day or darunavir/cobicistat 800/150 mg 1 cp / day), and hydroxychloroquine cp 200 mg, 1 cp x 2 / day.
  Interventions: Dietary Supplement: SivoMixx (200 billion); Drug: Azithromycin; Drug: hydroxychloroquine

INTERVENTIONS:
Dietary Supplement: SivoMixx (200 billion) — Composition of SivoMixx: Streptococcus thermophilus DSM322245, Bifidobacterium lactis DSM 32246, Bifidobacterium lactis DSM 32247, Lactobacillus acidophilus DSM 32241, Lactobacillus helveticus DSM 32242, Lactobacillus paracasei DSM 32243, Lactobacillus plantarum DSM 32244, Lactobacillus brevis DSM 27961 (NB: DSM n°... : bacterial strain identification code)
  Groups: bacteriotherapy
Drug: Azithromycin — dose: 500mg 1 cp / day (alternatively lopinavir/ritonavir cps 200/50 mg, 2 cps x 2 / day or darunavir 800 mg 1 cp / day + ritonavir 100 mg 1 cp / day or darunavir/cobicistat 800/150 mg 1 cp / day)
Drug: hydroxychloroquine — dose: 200 mg, 1 cp x 2 / day

SUMMARY:
In light of its high morbidity and mortality, COronaVIrus Disease 19 (COVID-19) pandemic spread is considered an unprecedented global health challenge.

Given the very limited therapeutic options available against Severe Acute Respiratory Syndrome - CoronaVirus-2 (SARS-CoV-2) epidemic at this time, the evaluation of new resources, designed in the first instance for other pathologies but potentially active against COVID-19, represents a priority in clinical research.

This is an observational, retrospective, non-profit study on the adjuvant use of bacteriotherapy in the early control of disease progression in patients affected by COVID-19 and treated with the current standard of care on the basis of the interim guidelines of the Italian Society of Infectious and Tropical Diseases.

The main purpose of the study is to evaluate the effectiveness of bacteriotherapy in reducing the clinical impact of acute diarrhea, containing the progression of COVID-19 and preventing the need for hospitalization in intensive care units.

DETAILED DESCRIPTION:
Italy was the first European country hit by the severe outbreak of the SARS-CoV-2 epidemic emerged from China, with a high morbidity and associated mortality.

Given the limited treatment options currently available, the search for resources capable of improving disease outcomes is fundamental for the management of patients

Systemic inflammation related to COVID-19, dietary changes, and use of antibiotics are all variables that contribute to changes in the gut microbiota with significant impact on the disease outcomes. Probiotic supplementation can help to correct these issues.

Moreover some strains of lactobacilli and bifidobacteria inhibit influenza virus, rhinovirus, respiratory syncytial virus, adenovirus, and pneumovirus .

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosis
* symptomatic COVID-19
* hospitalization in infectious diseases wards

Exclusion Criteria:

* Pregnant
* hospitalization in Intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients affected by COVID-19 admitted to Policlinico Umberto I, University of Rome "Sapienza" (Italy), between March 14, 2020 and April 4, 2020.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
delta of time of disappearance of acute diarrhea | 21 days
  Comparison between the two groups. Acute diarrhea was defined as a stool with increased water content, volume, or frequency that lasts less than 14 days.

SECONDARY OUTCOMES:
Delta in the number of patients requiring orotracheal intubation despite treatment | 21 days
  Comparison between the two groups
Delta of crude mortality | 21 days
  Comparison between the two groups
Delta of length of stay for patients in hospital | 21 days
  Comparison between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella d'Ettorre, MD, PhD, Principal Investigator — University of Rome Sapienza - Policlinico Umberto I Rome (Italy)
Locations (1):
- Department of Public Heath and Infectious Diseases. University of Rome "Sapienza" (Italy), Rome, Italy

REFERENCES:
- [Result] Patel R, DuPont HL. New approaches for bacteriotherapy: prebiotics, new-generation probiotics, and synbiotics. Clin Infect Dis. 2015 May 15;60 Suppl 2(Suppl 2):S108-21. doi: 10.1093/cid/civ177. PMID 25922396
- [Result] Jiang X, Hou X, Tang L, Jiang Y, Ma G, Li Y. A phase trial of the oral Lactobacillus casei vaccine polarizes Th2 cell immunity against transmissible gastroenteritis coronavirus infection. Appl Microbiol Biotechnol. 2016 Sep;100(17):7457-69. doi: 10.1007/s00253-016-7424-9. Epub 2016 Mar 28. PMID 27020282
- [Result] Jayawardena R, Sooriyaarachchi P, Chourdakis M, Jeewandara C, Ranasinghe P. Enhancing immunity in viral infections, with special emphasis on COVID-19: A review. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):367-382. doi: 10.1016/j.dsx.2020.04.015. Epub 2020 Apr 16. PMID 32334392